CLINICAL TRIAL: NCT03377400
Title: Phase II Trial of Durvalumab (MEDI4736 )/Tremelimumab Combined With Definitive Concurrent Chemo-radiotherapy for Inoperable Esophageal Squamous Cell Carcinoma
Brief Title: Definitive CCRT Combined With Durvalumab and Tremelimumab for Inoperable Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Mu Sun, Associated Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2017-06-138
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — durvalumab; tremelimumab; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): Concurrent radiotherapy with chemotherapy (5FU/CDDP) and immune checkpoint inhibitors (durvalumab/tremelimumab), and followed by consolidation immune checkpoint inhibitors
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — concurrent radiotherapy
  Other Names: tremelimumab; 5FU; Cisplatin

SUMMARY:
This is a single arm phase II study, in which 2 cycles of chemotherapy (5FU/CDDP) and immunotherapy (durvalumab and tremelimumab) are administered every 3 weeks with concurrent radiotherapy for inoperable locally advanced esophageal squamous cell carcinoma. Four weeks after completion of CCRT combined with immunotherapy, 2 cycles of durvaluma and tremelimumab will be administered every 4 weeks and thereafter durvalumab monotherapy Q4W will be maintained until unacceptable toxicity or disease progression, or for maximum 2 years after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous esophageal cancer
* The clinical stage T2-3N0M0 or T1-3N1-3M0
* Inoperable case: it refers to medically inoperable status and/or patient's refusal to surgery and/or cervical location and/or locoregionally recurrent tumor after primary surgery
* ECOG PS of 0 to 1

Exclusion Criteria:

* clinical T4 disease (for example, invasion to aorta, vertebral body, or trachea/bronchus) or distant metastasis (M1)
* previously received radiotherapy for esophageal cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 year
  Time interval from enrollment to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Mu Sun, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, MA, South Korea